CLINICAL TRIAL: NCT07076251
Title: Building Access to Food Through Systems and Solidarity (BASIS): A Subsidized and Culturally-adapted Produce Box Program for Immigrant Communities of Brooklyn, NY - Family Box Pilot Study
Brief Title: Building Access to Food Through Systems and Solidarity (BASIS): A Subsidized and Culturally-adapted Produce Box Program for Immigrant Communities of Brooklyn, NY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-01962; R01MD018204 (NIH)
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Cardiometabolic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chinese American families living in New York City (NYC) (Experimental): Participants will receive a box, once a month across one year for a total of 12 boxes, with culturally relevant ingredients, books, and educational materials.
  Interventions: Other: Family Box program

INTERVENTIONS:
Other: Family Box program — Boxes will include approximately five pounds of dry ingredients (e.g., whole grains, legumes, flour), which translates into about 40 servings of food for a family of four per month. Each ingredient box will include culturally relevant recipes and, six times out of the twelve boxes, include a culturally relevant book for the family's child/children.

SUMMARY:
The goal of this study is to improve diet and social cohesion among Chinese American families living in New York City (NYC) through a program that provides whole grains and legumes, builds ethnic identity, and fosters family resilience. The study ultimately aims to leverage this program to address cardiometabolic disease disparities in a culturally meaningful way.

DETAILED DESCRIPTION:
The goal of this study is to improve diet and social cohesion among Chinese American families living in New York City (NYC). In this 12-month program, families will receive a box of whole grains and legumes, bilingual children's books (every other month), and nutrition education/recipes every month. This project is a partnership between NYU and 3 multisectoral organizations (i.e., a local farm, community-based organization, and bilingual book subscription company). The program will be evaluated using surveys at the beginning and end of the 12-month program. Through this pre-post evaluation, the investigators will evaluate the impact of the program on intake of whole grains and fruits and vegetables (inclusive of legumes). The study ultimately aims to leverage this program to address cardiometabolic disease disparities in a culturally meaningful way.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-90 years
2. Self-identify as Chinese or Chinese American
3. Caretaker or parent of at least one child who lives with them between the ages of 2-6 years
4. Willing and able to provide written consent
5. Comfortable speaking English, Cantonese, or Mandarin; reading in English or simplified or traditional Chinese
6. Can travel to CPC site for box pick-up monthly

Exclusion Criteria:

1. Individuals who don't meet the eligibility criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in daily intake of whole grains (ounces/day) as assessed by the National Cancer Institute's (NCI) 26-item Dietary Screener Questionnaire (DSQ) | Baseline, End of Intervention (~12 months)
  The National Cancer Institute's (NCI) 26-item Dietary Screener Questionnaire (DSQ) is a tool used to assess dietary intake. It focuses on the frequency of consumption of specific foods and beverages within the past month. The DSQ is designed to capture intakes of fruits and vegetables, dairy/calcium, added sugars, whole grains/fiber, red meat, and processed meat.
Change in daily intake of fruits and vegetables (inclusive of legumes; cups/day) as assessed by the NCI 26-item DSQ | Baseline, End of Intervention (~12 months)
  The NCI 26-item DSQ is a tool used to assess dietary intake. It focuses on the frequency of consumption of specific foods and beverages within the past month. The DSQ is designed to capture intakes of fruits and vegetables, dairy/calcium, added sugars, whole grains/fiber, red meat, and processed meat.

SECONDARY OUTCOMES:
Change in Family functioning score | Baseline, End of Intervention (~12 months)
  Family functioning score will be assessed via self-report using a validated questionnaire about family interactions and dynamics.
Change in the percent of individuals who report that they have food insecurity | Baseline, End of Intervention (~12 months)
  Outcome measure is assessed through a self-administered survey.

CONTACTS AND LOCATIONS:
Overall Officials: Madison N LeCroy, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
De-identified IPD data will not be made available due to the following key reasons. First, the possibility of re-identification of participants if IPD were shared is more than minimal given the small sample size, community-based recruitment, and eligibility criteria. Participants have expressed heightened concerns about data security, and thus the study team will take efforts to protect participants by restricting access to their IPD. Secondly, data-sharing de-identified IPD is not included in the study's consent form, and re-consenting enrolled participants with this added stipulation would not be feasible.